CLINICAL TRIAL: NCT02053428
Title: Comparison of Percutaneous Image-guided Gastrostomies: A Single Centre Pilot Study
Brief Title: Comparison of Percutaneous Image-guided Gastrostomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0298B
Record Dates: First submitted 2014-01-21; First posted 2014-02-03 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-01

CONDITIONS: Cancer of Head and Neck
Keywords: Head and neck cancer; Percutaneous image-guided gastrostomy; Pain; Quality of life; Complication
MeSH Terms: conditions — Head and Neck Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastrostomy - pull technique (Active Comparator): Percutaneous image-guided gastrostomy using large-bore mushroom-retained catheters via the pull technique
  Interventions: Procedure: percutaneous image-guided gastrostomy
- Gastrostomy - push technique (Active Comparator): Percutaneous image-guided gastrostomy using small-bore cope loop catheters via the push technique
  Interventions: Procedure: percutaneous image-guided gastrostomy

INTERVENTIONS:
Procedure: percutaneous image-guided gastrostomy

SUMMARY:
Percutaneous image-guided gastrostomy (PIG) is an increasingly popular technique of creating gastroenteric access through the anterior abdominal wall for nutrition and/ or compression. Large-bore mushroom-retained catheters via the pull technique and small-bore cope loop catheters via the push technique are both used at Interventional Radiology for PIG at our institution. To date, there is no guideline for PIG and no direct comparison of two PIG techniques. The proposed pilot study is to compare the two different types of PIG techniques in head and neck cancer patients who require prophylactic enteral feeding by PIG. The purpose of the study is to assess the feasibility of a large randomized clinical trial to compare these two PIG techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years;
2. Life expectancy > 6 months;
3. Diagnosed with head and neck cancer; and
4. Scheduled to have prophylactic enteral feeding by percutaneous image-guided gastrostomy performed in the interventional radiology suite.

Exclusion Criteria:

1. Pregnancy; or
2. Established pharyngeal obstruction and/or presence of an enteral feeding device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pain experience | pre, 1-hour, 2-hour, 3-hour, 1-day, 2-day, 3-day and weekly for up to six weeks post procedure
  The primary objective of this study is to compare the level of pain experienced, measured by the dose of sedation used during the procedure, and numerical rating scale (NRS)

SECONDARY OUTCOMES:
Technical success | Day 0 post procedure
  successful placement of percutaneous image-guided gastrostomy
Catheter malfunction rate | Up to six months post procedure
  tube clogging, dislodgement and/or leakage
Tube site complications | Up to six months post procedure
  Skin infection on tube exit
Quality of life | Up to six weeks post procedure
  Quality of life for patients undergoing different types of PIG procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Kong Teng Tan, MB BCH BAO, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada